CLINICAL TRIAL: NCT06837441
Title: Atrial Fibrillation Termination Versus Prespecified Ablation for Persistent Atrial Fibrillation:A Pilot Study
Brief Title: PerAF: AF Termination vs Prespecified Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: The Shanghai Yangpu Central Hospital (Unknown); Jinshan Hospital Affiliated to Fudan University (Unknown)
Responsible Party: Principal Investigator, Xu Liu, Doctor Liu, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TPAF
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2023-01

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AF-termination group (Experimental)
  Interventions: Procedure: Atrial Fibrillation Termination
- Prespecified-ablation group (Sham Comparator)
  Interventions: Procedure: Prespecified Ablation

INTERVENTIONS:
Procedure: Atrial Fibrillation Termination — Pursuing Atrial Fibrillation Termination as a Procedural Endpoint
  Arms: AF-termination group
Procedure: Prespecified Ablation — Prespecified Ablation Strategy Followed by Cardioversion
  Arms: Prespecified-ablation group

SUMMARY:
The design of this study is an intervention, randomized, controlled study and contains two randomized groups：（1）AF-termination group；（2）Prespecified-ablation group.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18 and 80 years old;
2. Patients undergoing a first-time ablation procedure for PersAF, and in spontaneous AF at the beginning of the procedure;
3. Diagnosed as persistent AF according to the latest clinical guidelines，with atrial fibrillation lasting for at least one month;
4. Ineffective or intolerable to ≥1 anti-arrhythmia drug treatment;
5. Patients must be able and willing to provide written informed consent to participate in this study;
6. Patients must be willing and able to comply with all study follow- up requirements.

Exclusion Criteria:

1. .Uncontrolled congestive heart failure, EF <35%;
2. . History of severe valve disease and/or prosthetic valve replacement;
3. . Myocardial infarction or stroke within 6 months;
4. . Severe congenital heart disease;
5. . Left atrial diameter ≥60mm;
6. . Contrast agent allergy;
7. . The use of anticoagulant drugs is contraindicated;
8. . Severe lung disease;
9. . Left atrial thrombus confirmed by preoperative esophageal ultrasound;
10. .Contraindications for cardiac catheterization;
11. .Prior left atrial ablation (surgical or catheter);
12. .Have performed any cardiac surgery within 2 months;
13. .Poor general health;
14. .Life expectancy < 12 months, including factors such as physical inability to tolerate ablation or unstable disease conditions.-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Freedom from any documented atrial arrhythmia - atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL) - of more than 30 seconds, excluding the initial 3 months blanking period, at a minimum of 12 months follow up after a single ablat | 12 months

SECONDARY OUTCOMES:
Freedom from AF after a single procedure without anti-arrhythmic medications (excludes the blanking period) at 12 months； | 12 months
Freedom from AF/AT/AFL after a single procedure with/without anti-arrhythmic medications (excludes the blanking period) at 12 months | 12 months
Freedom from AF after a single procedure with/without anti-arrhythmic medications (excludes the blanking period) at 12 months | 12 months
Freedom from any AT episodes lasting more than 30 seconds after the blanking period without AADs after a single procedure | 12 months
Incidence of periprocedural adverse events. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No